CLINICAL TRIAL: NCT02169089
Title: Mineralocorticoid Receptor Antagonism Clinical Evaluation in Atherosclerosis Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: University of Maryland (Other); University of Toronto (Other); Winthrop University (Other)
Responsible Party: Principal Investigator, Sanjay Rajagopalan, Chief, Cardiovascular Medicine, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 57047
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spironolactone (Experimental): Spironolactone
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — Patients will be given Spironolactone 12.5 mg on week 0 (visit 2). Patients will be escalated to 25 mg daily Spironolactone or maximal tolerated dose over a 4-week period. Patients will continue treatment for an additional 48 weeks.
  Other Names: Aldactone
  Arms: Spironolactone
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Atherosclerotic disease, or hardening of the arteries, is characterized by the thickening of the arterial walls due to fatty deposits in wall and inflammation in the wall of arteries. High cholesterol, high blood pressure, diabetes, obesity and genetics play an important role in developing clinical symptoms of atherosclerosis disease. The complications of advanced atherosclerosis are chronic, slowly progressive and cumulative, resulting in heart attack, stroke and/or death and blockage of arteries.

This study is being done to assess the effectiveness of Spironolactone therapy to slow down the worsening of atherosclerotic disease (hardening of the arteries) in aorta (this is a large vessel coming out of your heart) compared to placebo (look alike sugar pill). This will be checked by comparing before and after therapy magnetic resonance imaging (MRI) pictures of your aortic wall.

Spironolactone is an FDA approved drug used to treat heart failure and in the management of hypertension (high blood pressure), but in this study it is used for another unapproved reason. In this study, we would like to evaluate the effects of Spironolactone in people with diabetes and atherosclerotic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients >45 or >40 years with known atherosclerotic events (examples include MI, Stroke) and able to provide informed consent (females must be either post-menopausal for one year, surgically sterile, or using effective contraception. Oral contraceptives are disallowed.
2. Patients with Type II Diabetes with HbA1c ≤ 9.0 on stable anti-glycemic regimen that may include oral and/or injectable therapy (GLP-1/Insulin etc.). Changes in dose of glycemic regimen is allowed during the course of the trial if felt to be clinically appropriate.
3. GFR <90 and evidence of proteinuria (Urine albumin/creatinine ratio of >30 mg/g or equivalent) in a urine specimen within 12 months OR GFR <60 mg/g regardless of proteinuria.
4. Patients must be on ACE and/or ARB therapy with no planned dose adjustments.

Exclusion Criteria:

1. Uncontrolled hypertension (SBP>160 and/or DBP>95 mmHg at visit 0 (screening) and SBP >145 mm Hg at visit 2).
2. GFR (MDRD) of <15 at Visit 0 (screening).
3. Hyperkalemia defined as serum K+≥ 5.1 meq/L at visit 0 (screening).
4. LDL cholesterol >150 mg/dl.
5. Plasma triglycerides >400 mg/dl.
6. Contraindications to MRI (metallic implants, severe claustrophobia).
7. Acute coronary syndrome, Transient ischemic attack, CVA or critical limb ischemia during the last 6 months or coronary/peripheral revascularization within the last 3 months.
8. Evidence of a secondary form of hypertension.
9. Initiation of new therapy with statins, ACEI/ARB, anti-oxidants, CCBs, diuretics, β blockers.
10. Type I diabetes mellitus
11. Known contraindication, including history of allergy to Spironolactone.
12. . Any surgical or medical condition which might alter pharmacokinetics of drug (e.g. renal transplant, liver failure, liver transplant).
13. Concurrent potentially life threatening arrhythmia or symptomatic arrhythmia.
14. Significant hyponatremia defined as Na <130 meq/L.
15. History of prior malignancy including leukemia and lymphoma (but not basal cell skin cancer, cured squamous cell cancer and localized Prostate cancer).
16. History of any severe, life-threatening disease.
17. Any surgical or medical conditions which places the patient at higher risk derived from his/her participation into the study, or likely to prevent patient from complying with requirements.
18. History of drug abuse within the last 2 years, noncompliance and unwillingness/inability to consent.
19. Pregnant women and nursing mothers.
20. Class III or IV Congestive Heart Failure.
21. Primary Hyperaldosteronism.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Rajagopalan, Principal Investigator — Chief, Cardiovascular Medicine
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Rajagopalan S, Dobre M, Dazard JE, Vergara-Martel A, Connelly K, Farkouh ME, Gaztanaga J, Conger H, Dever A, Razavi-Nematollahi L, Fares A, Pereira G, Edwards-Glenn J, Cameron M, Cameron C, Al-Kindi S, Brook RD, Pitt B, Weir M. Mineralocorticoid Receptor Antagonism Prevents Aortic Plaque Progression and Reduces Left Ventricular Mass and Fibrosis in Patients With Type 2 Diabetes and Chronic Kidney Disease: The MAGMA Trial. Circulation. 2024 Aug 27;150(9):663-676. doi: 10.1161/CIRCULATIONAHA.123.067620. Epub 2024 Aug 12. PMID 39129649

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spironolactone | Placebo
Started | 37 | 42
Completed | 26 | 25
Not Completed | 11 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spironolactone | Placebo | Total
Number analyzed (Participants) | 37 | 42 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (8.3) | 63.2 (8.7) | 64.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 21 | 25 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 26 | 46
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Atheroma Volume (PAV) in the Thoracic Aorta of Spironolactone vs. Placebo
Time Frame: 56 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 37 | 42
percentage change | 0.5 (10.3) | 7.3 (11.4)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.0293, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -7.78

2. Secondary Outcome: Left Ventricular Mass Index of Spironolactone vs. Placebo.
Time Frame: 56 weeks
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 37 | 42
g/m^2 | -3.5 (3.7) | 2.1 (4.5)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -2.6 — The mean reported -3.5 and 2.1 represents the mean change between follow-up & baseline visit. The statistical test (Mann-Whitney) reported Median difference of -2.6, which corresponds to the difference between the spironolactone and placebo group

3. Secondary Outcome: Myocardial Fibrosis (Change in Native T1) Spironolactone vs. Placebo
Time Frame: 56 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 37 | 42
ms | -10.3 (35.9) | 17.1 (35.6)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.0189, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -40.7 — The mean reported -10.3 and 17.1 represents the mean change between follow-up & baseline visit. The statistical test (Mann-Whitney) reported Median difference of -2.6, which corresponds to the difference between the spironolactone and placebo group

4. Secondary Outcome: Change in 24-hour Ambulatory Systolic Blood Pressure of Spironolactone vs. Placebo
Time Frame: 11 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 37 | 42
mmHg | -5.95 (10.9) | 2 (17.59)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.1276, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -7.5 — The mean reported -5.95 and 2 represents the mean change between follow-up & baseline visit. The statistical test (Mann-Whitney) reported Median difference of -2.6, which corresponds to the difference between the spironolactone and placebo group

5. Secondary Outcome: Measures of Insulin Resistance (HOMA-IR) of Spironolactone vs. Placebo
Time Frame: 56 weeks
Population: Data not collected for this outcome measure.
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: AEs were monitored by blood work, self report, vital signs, and MRI.
Arm/Group | Spironolactone | Placebo
All-Cause Mortality (participants affected / at risk) | 1/37 | 1/42
Serious Adverse Events (participants affected / at risk) | 7/37 | 8/42
Other Adverse Events (participants affected / at risk) | 9/37 | 8/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spironolactone (N=37) | Placebo (N=42)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diabetes related (Endocrine disorders) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 2 (2)
Surgical (Surgical and medical procedures) | 1 (1) | 4 (4)
Chest pain/discomfort (Cardiac disorders) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spironolactone (N=37) | Placebo (N=42)
Hyperkalemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Diabetes related (Endocrine disorders) | 2 (2) | 2 (2)
Hypotension (Cardiac disorders) | 3 (3) | 1 (1)
AKI (Renal and urinary disorders) | 0 (0) | 1 (1)
Chest pain/discomfort (Cardiac disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)
Neck spasms (General disorders) | 0 (0) | 1 (1)
Breast tenderness/Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT02169089/Prot_SAP_000.pdf